CLINICAL TRIAL: NCT00573352
Title: Phase 1 Study to Determine the Efficacy of Using Energy Specific Far Infrared (FIR) Radiation for the Treatment of Arthritis and Other Related Diseases
Brief Title: Far Infrared Radiation Treatment for Osteoarthritis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GAAD Medical Research Institute Inc. (Other)
Responsible Party: Dr. Kwasi Donyina, GAAD Medical Research Institute Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAAD-OA-CTP1
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2009-01-05 (Estimated); Status verified 2009-01

CONDITIONS: Osteoarthritis
Keywords: Arthritis, Degenerative; Osteoarthrosis; Osteoarthrosis Deformans
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Far infrared radiation
  Interventions: Radiation: Far Infrared

INTERVENTIONS:
Radiation: Far Infrared — Far Infrared Radiation (5μm to 20μm wavelength). Duration is 30 to 40 minutes per session

SUMMARY:
A study to evaluate the possibility of using far infrared radiation to manage pain due to osteoarthritis.

DETAILED DESCRIPTION:
Arthritis consists of more than 100 different conditions. These conditions range from relatively mild forms such as tendonitis and bursitis to crippling forms as rheumatoid arthritis. Pain syndromes include fibromyalgia and arthritis-related disorders as lupus erythematosus that involve every part of the body. There are forms of the disease, such as gout that almost nobody connects with arthritis. Osteoarthritis is the most common form of arthritis.

The objective for the study is to access the possibility of using far infrared radiation for pain management.

ELIGIBILITY:
Inclusion Criteria:

* 1 year old and above

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2006-09; Primary Completion 2008-02 (Actual); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
The primary end point is to determine the therapeutic effects of far infrared radiation on osteoarthritis | 2 years and 9 months

SECONDARY OUTCOMES:
The therapeutic effects of far infrared radiation on all forms of arthritis | 2 years and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Kwasi Donyina, Ph.D., Study Director — GAAD Medical Research Institute Inc.; Ken Nedd, M.D., Principal Investigator — GAAD Medical Research Institute Inc.
Locations (1):
- The Centre for Incurable Diseases, Toronto, Ontario, Canada